CLINICAL TRIAL: NCT05872321
Title: Assessment of the New Lateral Sinus Floor Elevation Technique Using Piezosurgery: A Clinical and Radiographic Prospective Study
Status: Completed | Type: Observational
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Christian Makary, Professor, Saint-Joseph University
Other Study IDs: FMD-SF86
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2023-06

CONDITIONS: Lateral Sinus Lift; Per-operation Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Per-operative Complication
  Interventions: Other: Complication

INTERVENTIONS:
Other: Complication — whether or not complications occur

SUMMARY:
For patients requiring LSFE, demographic data, including age, sex and smoking habits were collected. Preoperative CBCT images were analyzed for radiographic assessment of risk factors through measurement of sinus mucosa thickness, sinus lateral wall thickness, sinus width, presence of Underwood's septa, and presence of the alveolar antral artery. A bone consuming technique using piezosurgery was implemented. This technique involved eroding the buccal bone prior to window outlining followed mucosal elevation using novel ultrasonic curettes. sinus mucosa perforation, hemorrhage, and postoperative infectious complications were documented. The measurement of the studied factors was performed on Newtom VGI viewer software, by two evaluators J.B. and A.M.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received lateral sinus floor elevation using this new piezosurgery technique.

Exclusion Criteria:

* the usual exclsion criteria for external sinus lift procedure

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the patient needing lateral sinus lift procedure prior to implant placement.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Perioperative complication | During surgical procedure
  We will monitor the prevalence of membrane perforation during external sinus lift procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided